CLINICAL TRIAL: NCT06487845
Title: Single and Multiple Dose Escalation Study to Investigate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BAY 3283142 Given as Immediate Release (IR) Tablets in Chinese Healthy Participants in a Randomized, Placebo-controlled, Single-blind, Group-comparison Design
Brief Title: A Study to Learn How Safe BAY3283142 is When Taken as a Single Dose or as Multiple Doses in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22420
Record Dates: First submitted 2024-06-24; First posted 2024-07-05 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Chronic Kidney Disease; Non-proliferative Diabetic Retinopathy; Healthy Volunteers
Keywords: CKD; NPDR
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose step 1 (Experimental): Participants will receive a low dose of BAY3283142 on Day 1 followed by 1 day without dosing and a multiple dose phase for 7 days.
  Interventions: Drug: BAY3283142
- Dose step 2 (Experimental): Participants will receive a high dose of BAY3283142 on Day 1 followed by 1 day without dosing and a multiple dose phase for 7 days.
  Interventions: Drug: BAY3283142
- Placebo (Placebo Comparator): Participants will receive placebo on Day 1 followed by 1 day without dosing and a multiple dose phase for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY3283142 — IR tablets, oral
  Arms: Dose step 1; Dose step 2
Drug: Placebo — Placebo matched to BAY3283142
  Arms: Placebo

SUMMARY:
Researchers are looking for a better way to treat people who have chronic kidney disease (CKD) or non-proliferative diabetes retinopathy (NPDR). CKD is a long-term condition in which the ability of the kidneys to work decreases over time. It is often caused by high blood glucose levels. NPDR is another condition in which high blood glucose levels cause damage to the blood vessels of the retina, which is a tissue at the back of the eyes.

The study drug BAY3283142 works by activating a protein called soluble guanylate cyclase, which helps widen the blood vessels and regulate blood flow inside the body. This may help increase the blood flow in the kidneys and improve their function. It could also help to restore blood flow to the retina.

This study will include healthy participants who will not benefit from taking BAY3283142. However, the study will provide information on how to test BAY3283142 in future studies in participants with CKD or NPDR.

The main purpose of this study is to check how safe single and multiple doses of BAY3283142 are in healthy Chinese participants.

For this, researchers will collect the number and percentage of participants who have medical problems, which are also known as 'adverse events', after taking BAY3283142 or a placebo. A placebo looks like the study treatment but does not have any medicine in it.

The study doctor will keep track of all adverse events that happen in the study, even if they are not related to the study treatments.

The participants will be randomly divided into 2 treatment groups. They will take either BAY3283142 as an immediate-release tablet, or a placebo tablet, once, by mouth, based on the group assigned to them. An immediate-release tablet quickly dissolves and releases the drug inside the body.

Participants will have a one-day break after taking the single dose and then continue taking their assigned treatment once daily for a week. Researchers will check two different dose strengths of BAY3283142 in this study, starting with a low dose first.

Each participant will be in the study for around 7 weeks, which includes:

A visit within 21 days before the first dose to confirm if the participant can take part in the study

A hospital stay of 15 days during which the participant will take the assigned study treatment and the study doctor will monitor the participant's health

A visit after 7 to 10 days of taking the last dose during which the study doctor will perform a health check-up of the participant

During the study, the study doctor and his/her team will:

Test participants' blood and urine samples and check their overall health

Monitor participants' heart health by electrocardiogram (ECG) and measure their blood pressure and heart rate

As this study is conducted in healthy participants who will not gain any benefit from the treatment, access to the treatment after the study is not planned.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 to 45 years of age (both inclusive) at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory test and 12-lead ECG.
* Race: Chinese
* Body mass index (BMI) within the range 18.0 - 27.9 kg/m² (both inclusive) at screening.
* Body weight of at least 55 kg at screening.
* Male and female, female only allowed in the 5 mg dose group. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Known tendency for vasovagal reactions (e.g., after venipuncture) or history of syncope.
* Systolic blood pressure below 100 mmHg or above 140 mmHg (after 15 minutes of supine rest) at screening.
* Diastolic blood pressure below 60 mmHg or above 90 mmHg (after 15 minutes of supine rest) at screening.
* Heart rate below 50 or above 90 beats per minute (after 15 minutes of supine rest) at screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-04 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse event (TEAEs) | From first study intervention administration until [including] 7 days after end of treatment with study intervention (approximately 25 days)
Percentage of participants with treatment emergent adverse event (TEAEs) | From first study intervention administration until [including] 7 days after end of treatment with study intervention (approximately 25 days)

SECONDARY OUTCOMES:
AUC of BAY3283142 | 0 to 48 hours post-dose after the first dose on Day 1
  AUC: Area under the concentration vs. Time curve from zero to infinity after single (first) dose
Cmax of BAY3283142 | 0 to 48 hours post-dose after the first dose on Day 1
  Cmax: Maximum observed drug concentration in measured matrix after single dose administration, directly taken from analytical data
AUC/D of BAY3283142 | 0 to 48 hours post-dose after the first dose on Day 1
  AUC/D: AUC divided by dose
Cmax/D of BAY3283142 | 0 to 48 hours post-dose after the first dose on Day 1
  Cmax/D: Cmax devided by dose
AUCτ,md of BAY3283142 | 0 to 24 hours post-dose after the last dose on Day 9
  AUCτ,md: AUC during any dose interval after multiple dose
Cmax,md of BAY3283142 | 0 to 24 hours post-dose after the last dose on Day 9
  Cmax,md: Maximum observed drug concentration in measured matrix after multiple dose administration during a dosage interval, directly taken from analytical data
AUCτ,md/D of BAY3283142 | 0 to 24 hours post-dose after the last dose on Day 9
  AUCτ,md/D: AUC during any dose interval after multiple dose divided by dose
Cmax,md/D of BAY3283142 | 0 to 24 hours post-dose after the last dose on Day 9
  Cmax,md/D: Cmax,md divided by dose

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou University of TCM, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.